CLINICAL TRIAL: NCT00734604
Title: A Comparison of Psychosocial Outcomes Following Tadalafil Once a Day or PDE5 Inhibitor As Needed in Men With Erectile Dysfunction.
Brief Title: A Study for Patients With Erectile Dysfunction to Test Whether Tadalafil Taken Once a Day Can Better Improve Psychological Outcomes.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12313; H6D-CR-S024 (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Results first posted 2010-11-18 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-10

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil; Sildenafil Citrate; Health Services Needs and Demand

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- T(OaD)/S(PRN)/T(PRN) (Experimental): Tadalafil 5 mg once a day [T(OaD)] for 8 weeks, 1 week washout, sildenafil citrate 100 mg as needed [S(PRN)] for 8 weeks, 1 week washout, tadalafil 20 mg as needed [T(PRN)] for 8 weeks
  Interventions: Drug: tadalafil once a day [T(OaD)]; Drug: sildenafil citrate as needed [S(PRN)]; Drug: tadalafil as needed [T(PRN)]
- T(OaD)/T(PRN)/S(PRN) (Experimental): Tadalafil 5 mg once a day [T(OaD)] for 8 weeks, 1 week washout, tadalafil 20 mg as needed [T(PRN)] for 8 weeks, 1 week washout, sildenafil citrate 100 mg as needed [S(PRN)] for 8 weeks
  Interventions: Drug: tadalafil once a day [T(OaD)]; Drug: sildenafil citrate as needed [S(PRN)]; Drug: tadalafil as needed [T(PRN)]
- S(PRN)/T(OaD)/T(PRN) (Experimental): Sildenafil citrate 100 mg as needed [S(PRN)] for 8 weeks, 1 week washout, tadalafil 5 mg once a day [T(OaD)] for 8 weeks, 1 week washout, tadalafil 20 mg as needed [T(PRN)] for 8 weeks
  Interventions: Drug: tadalafil once a day [T(OaD)]; Drug: sildenafil citrate as needed [S(PRN)]; Drug: tadalafil as needed [T(PRN)]
- S(PRN)/T(PRN)/T(OaD) (Experimental): Sildenafil citrate 100 mg as needed [S(PRN)] for 8 weeks, 1 week washout, tadalafil 20 mg as needed [T(PRN)] for 8 weeks, 1 week washout, tadalafil 5 mg once a day [T(OaD)] for 8 weeks
  Interventions: Drug: tadalafil once a day [T(OaD)]; Drug: sildenafil citrate as needed [S(PRN)]; Drug: tadalafil as needed [T(PRN)]
- T(PRN)/T(OaD)/S(PRN) (Experimental): Tadalafil 20 mg as needed [T(PRN)] for 8 weeks, 1 week washout, tadalafil 5 mg once a day [T(OaD)] for 8 weeks, 1 week washout, sildenafil citrate 100 mg as needed [S(PRN)] for 8 weeks
  Interventions: Drug: tadalafil once a day [T(OaD)]; Drug: sildenafil citrate as needed [S(PRN)]; Drug: tadalafil as needed [T(PRN)]
- T(PRN)/S(PRN)/T(OaD) (Experimental): Tadalafil 20 mg as needed [T(PRN)] for 8 weeks, 1 week washout, sildenafil citrate 100 mg as needed [S(PRN)] for 8 weeks, 1 week washout, tadalafil 5 mg once a day [T(OaD)] for 8 weeks
  Interventions: Drug: tadalafil once a day [T(OaD)]; Drug: sildenafil citrate as needed [S(PRN)]; Drug: tadalafil as needed [T(PRN)]

INTERVENTIONS:
Drug: tadalafil once a day [T(OaD)] — 5 mg tablet taken once a day (OaD) by mouth for 8 weeks
  Other Names: Cialis; LY450190
Drug: sildenafil citrate as needed [S(PRN)] — 100 mg tablet taken as needed (PRN) by mouth for 8 weeks
Drug: tadalafil as needed [T(PRN)] — 20 mg tablet taken as needed (PRN) by mouth for 8 weeks
  Other Names: Cialis; LY450190

SUMMARY:
The primary purpose of the study is to help answer whether tadalafil taken once a day can help improve the psychological outcomes (such as sexual self confidence, spontaneity and time concerns) compared to sildenafil taken as needed in patients with erectile dysfunction (ED).

ELIGIBILITY:
Inclusion Criteria:

* History of erectile dysfunction (ED).
* Have had satisfactory response to tadalafil, sildenafil citrate, or vardenafil HCl for a period of at least 6 months and expect frequent use (at least one dose per week, on average) when administered as needed.
* Have never used tadalafil 5 mg or 2.5 mg once a day therapy.
* Anticipate having the same adult female sexual partner willing to participate during the study.
* Agree to make at least four sexual intercourse attempts during the first four weeks of the study.
* Agree not to use any other treatment for ED (even herbal treatments) during the study.
* Agree to follow the directions given by the study doctor and staff about using the study drug.

Exclusion Criteria:

* Have any other primary sexual disorders present or penile deformity.
* Have history of radical prostatectomy or penile implant.
* Have problems with your kidneys, liver, or nervous system.
* Have uncontrolled diabetes, as measured by a blood test for haemoglobin A1C greater than a value of 11%.
* Are being treated for heart disease with any drug that is called a nitrate (for example, nitroglycerin).
* Have chest pain (called unstable angina or angina) that requires treatment.
* Have heart disease that causes symptoms after you exert yourself.
* Have had any of the following in the past 90 days: Heart attack, also known as a myocardial infarction (MI); Heart bypass surgery (called coronary artery bypass graft surgery); Had a procedure to open up blood vessels in the heart known as angioplasty or stent placement (percutaneous coronary intervention).
* Have a history of loss of vision in one eye because of nonarteritic anterior ischemic optic neuropathy (NAION).
* Have retinitis pigmentosa.
* Have history of human immunodeficiency virus (HIV).
* Have very high or very low blood pressure (your study doctor will discuss the limits with you).
* Have had a stroke or a significant injury to your brain or spinal cord within the last 6 months.
* Have rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption Lactose intolerance.
* Have a scheduled or planned surgery requiring anaesthesia during the course of the study.
* Have a scheduled cataract surgery during the curse of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Easter Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (37):
- United States (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newport Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middlebury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plantation, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Federal Way, Washington
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adelaide, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malvern, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands, Western Australia
- Brazil (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goiânia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio Claro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sao Jose Rio Preto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Germany (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augsburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sassari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Joya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santurce
- Spain (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., A Coruña
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vigo
- United Kingdom (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, County Durham
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plymouth, Devonshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lichfield, Staffordshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London

REFERENCES:
- [Derived] Rubio-Aurioles E, Porst H, Kim ED, Montorsi F, Hackett G, Morales AM, Stuckey B, Buttner H, West TM, Huynh NN, Lenero E, Burns P, Kopernicky V. A randomized open-label trial with a crossover comparison of sexual self-confidence and other treatment outcomes following tadalafil once a day vs. tadalafil or sildenafil on-demand in men with erectile dysfunction. J Sex Med. 2012 May;9(5):1418-29. doi: 10.1111/j.1743-6109.2012.02667.x. Epub 2012 Mar 16. PMID 22429760

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T(OaD)/S(PRN)/T(PRN) | T(OaD)/T(PRN)/S(PRN) | S(PRN)/T(OaD)/T(PRN) | S(PRN)/T(PRN)/T(OaD) | T(PRN)/T(OaD)/S(PRN) | T(PRN)/S(PRN)/T(OaD)
Started | 62 | 63 | 63 | 63 | 63 | 64
Completed | 59 | 51 | 57 | 54 | 55 | 58
Not Completed | 3 | 12 | 6 | 9 | 8 | 6
Not completed — Adverse Event | 0 | 2 | 0 | 2 | 1 | 1
Not completed — Serious Adverse Event | 1 | 0 | 1 | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 2 | 2 | 4 | 2 | 3
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 2 | 0 | 0 | 1 | 0
Not completed — Sponsor Decision | 1 | 2 | 1 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1 | 2 | 1
Not completed — Lack of Efficacy | 0 | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T(OaD)/S(PRN)/T(PRN) | T(OaD)/T(PRN)/S(PRN) | S(PRN)/T(OaD)/T(PRN) | S(PRN)/T(PRN)/T(OaD) | T(PRN)/T(OaD)/S(PRN) | T(PRN)/S(PRN)/T(OaD) | Total
Number analyzed (Participants) | 62 | 63 | 63 | 63 | 63 | 64 | 378
Age Continuous [Mean (Standard Deviation); unit: years] | 58.53 (11.62) | 55.12 (8.89) | 55.40 (11.70) | 54.87 (12.04) | 59.04 (10.56) | 54.36 (10.28) | 56.21 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 62 | 63 | 63 | 63 | 63 | 64 | 378
Race/Ethnicity, Customized [Number; unit: participants]
  African | 1 | 1 | 1 | 4 | 3 | 2 | 12
  Caucasian | 41 | 44 | 46 | 41 | 43 | 40 | 255
  East Asian | 1 | 0 | 1 | 0 | 0 | 1 | 3
  Hispanic | 19 | 17 | 15 | 18 | 17 | 19 | 105
  Native American | 0 | 0 | 0 | 0 | 0 | 2 | 2
  West Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Australia | 3 | 4 | 5 | 4 | 4 | 4 | 24
  Germany | 7 | 6 | 6 | 7 | 7 | 7 | 40
  Italy | 5 | 5 | 4 | 6 | 4 | 5 | 29
  Mexico | 14 | 14 | 14 | 14 | 14 | 14 | 84
  Spain | 10 | 10 | 10 | 9 | 9 | 9 | 57
  United Kingdom | 6 | 8 | 7 | 7 | 8 | 8 | 44
  United States | 17 | 16 | 17 | 16 | 17 | 17 | 100
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m^2) | 28.35 (4.18) | 27.62 (2.65) | 27.77 (3.71) | 28.68 (4.74) | 27.80 (3.51) | 29.08 (4.26) | 28.22 (3.91)
Erectile Dysfunction (ED) Duration [Number; unit: participants]
  => 1 year | 59 | 61 | 58 | 58 | 61 | 59 | 356
  => than 6 months through <1 year | 3 | 2 | 5 | 5 | 2 | 5 | 22
ED Etiology [Number; unit: participants]
  Mixed | 25 | 26 | 21 | 23 | 23 | 28 | 146
  Organic | 22 | 28 | 29 | 29 | 30 | 25 | 163
  Psychogenic | 5 | 3 | 9 | 9 | 1 | 7 | 34
  Unknown | 10 | 6 | 4 | 2 | 9 | 4 | 35
Prior sildenafil citrate use as needed (PRN) [Number; unit: participants]
  Yes | 36 | 40 | 40 | 39 | 39 | 35 | 229
  No | 26 | 23 | 23 | 24 | 24 | 29 | 149
Prior Vardenafil HCl use [Number; unit: participants]
  Yes | 21 | 18 | 17 | 10 | 19 | 19 | 104
  No | 41 | 45 | 46 | 53 | 44 | 45 | 274

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Between Tadalafil Once a Day (OaD) and Sildenafil as Needed (PRN) in Sexual Self-Confidence Domain of Psychological and Interpersonal Relationship Scales (PAIRS)
Description: The PAIRS is a self-administed scale that assesses the broader psychological and interpersonal outcomes associated with erectile dysfunction and its treatment. Sexual Self-Confidence score is the average of responses on 6 PAIRS item scores. Sexual Self-Confidence scores range from 1 (strongly disagree) to 4 (strongly agree). Higher scores are indicative of greater sexual self-confidence.
Time Frame: baseline, 8 weeks of each treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tadalafil Once a Day [T(OaD)]: Tadalafil 5 mg once a day [T(OaD)]
- Sildenafil as Needed [S(PRN)]: Sildenafil citrate 100 mg as needed [S(PRN)]
Arm/Group | Tadalafil Once a Day [T(OaD)] | Sildenafil as Needed [S(PRN)]
Number analyzed (Participants) | 351 | 347
units on a scale
  Baseline | 2.24 (0.62) | 2.23 (0.63)
  Change from Baseline | 0.50 (0.78) [0.41 to 0.57] | 0.39 (0.67) [0.29 to 0.45]
Statistical Analysis 1: Comparison: Tadalafil Once a Day [T(OaD)] vs Sildenafil as Needed [S(PRN)]; Test type: Superiority or Other; p = 0.001, t-test — p-value is for difference in LS Means change from baseline between tadalafil OaD and Sildenafil PRN; Kenward-Roger approximation was used for denominator degrees of freedom in the mixed model; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [0.04 to 0.19], Standard Error of Mean 0.04

2. Secondary Outcome: Change From Baseline Between Tadalafil Once a Day (OaD) and Tadalafil as Needed (PRN) in Sexual Self-Confidence Domain of Psychological and Interpersonal Relationship Scales (PAIRS)
Description: as for outcome 1
Time Frame: baseline, 8 weeks of each treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tadalafil as Needed [T(PRN)]: Tadalafil 20 mg as needed [T(PRN)]
Arm/Group | Tadalafil Once a Day [T(OaD)] | Tadalafil as Needed [T(PRN)]
Number analyzed (Participants) | 351 | 354
units on a scale
  Baseline | 2.24 (0.62) | 2.24 (0.63)
  Change from Baseline | 0.50 (0.78) | 0.50 (0.72)
Statistical Analysis 1: Comparison: Tadalafil Once a Day [T(OaD)] vs Tadalafil as Needed [T(PRN)]; Test type: Superiority or Other; p = 0.872, t-test — p-value is for difference in Pairs Sexual Self-Confidence Domain Score LS Mean and Change from Baseline between Tadalafil OaD and Tadalafil PRN Population; Kenward-Roger approximation was used for denominator degrees of freedom in the mixed model; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.06 to 0.08], Standard Error of Mean 0.04 — LS Mean difference = Tadalafil OaD-Tadalafil PRN

3. Secondary Outcome: Change From Baseline to Endpoint in the Spontaneity Domain of PAIRS
Description: The PAIRS is a self-administed scale that assesses the broader psychological and interpersonal outcomes associated with erectile dysfunction and its treatment. Spontaneity score is the average of responses on 9 PAIRS item scores. Spontaneity scores range from 1 (strongly disagree) to 4 (strongly agree). Higher scores are indicative of greater spontaneity.
Time Frame: baseline, 8 weeks of each treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil Once a Day [T(OaD)] | Sildenafil as Needed [S(PRN)] | Tadalafil as Needed [T(PRN)]
Number analyzed (Participants) | 351 | 347 | 354
units on a scale
  Baseline | 3.06 (0.48) | 3.07 (0.48) | 3.07 (0.48)
  Change from Baseline | 0.10 (0.50) | -0.05 (0.49) | 0.07 (0.49)
Statistical Analysis 1: Comparison: Tadalafil Once a Day [T(OaD)] vs Sildenafil as Needed [S(PRN)]; Test type: Superiority or Other; p < 0.001, t-test — p-value is for difference between Tadalafil OaD and Sildenafil PRN change from baseline in LS Mean; Kenward-Roger approximation was used for denominator degrees of freedom in the mixed model; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0.10 to 0.20], Standard Error of Mean 0.03
Statistical Analysis 2: Comparison: Tadalafil Once a Day [T(OaD)] vs Tadalafil as Needed [T(PRN)]; Test type: Superiority or Other; p = 0.395, t-test — p-value is for difference between Tadalafil OaD and Tadalafil PRN in change from baseline in LS Mean; Kenward-Roger approximation was used for denominator degrees of freedom in the mixed model; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.03 to 0.07], Standard Error of Mean 0.03

4. Secondary Outcome: Change From Baseline to Endpoint in the Time Concerns Domain of PAIRS
Description: The PAIRS is a self-administed scale that assesses the broader psychological and interpersonal outcomes associated with erectile dysfunction and its treatment. Time Concerns score is the average of responses on 8 PAIRS item scores. Time Concerns scores range from 1 (strongly disagree) to 4 (strongly agree). Higher scores are indicative of greater sexual self-confidence.
Time Frame: baseline, 8 weeks of each treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil Once a Day [T(OaD)] | Sildenafil as Needed [S(PRN)] | Tadalafil as Needed [T(PRN)]
Number analyzed (Participants) | 351 | 347 | 354
units on a scale
  Baseline | 2.43 (0.53) | 2.42 (0.54) | 2.42 (0.53)
  Change from Baseline | -0.30 (0.03) | 0.00 (0.53) | -0.17 (0.55)
Statistical Analysis 1: Comparison: Tadalafil Once a Day [T(OaD)] vs Sildenafil as Needed [S(PRN)]; Test type: Superiority or Other; p < 0.001, t-test — p-value is for the difference between Tadalafil OaD and Sildenafil PRN in Change from Baseline in LS Mean; Kenward-Roger approximation was used for denominator degrees of freedom in the mixed model; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.36 to -0.25], Standard Error of Mean 0.03
Statistical Analysis 2: Comparison: Tadalafil Once a Day [T(OaD)] vs Tadalafil as Needed [T(PRN)]; Test type: Superiority or Other; p < 0.001, t-test — p-value is for the difference between Tadalafil OaD and Tadalafil PRN in Change from Baseline in LS Mean; Kenward-Roger approximation was used for denominator degrees of freedom in the mixed model; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.20 to -0.08], Standard Error of Mean 0.03

5. Secondary Outcome: Change From Baseline to Endpoint in the Erectile Function Domain of the International Index of Erectile Function (IIEF)
Description: Self-reported erectile function over the past 4 weeks. Scores range from 0 (low or no erectile function) to 5 (high erectile function) on 6 questions (1-5, 15 of the IIEF). Total Erectile Function Domain scores range from 0 to 30.
Time Frame: baseline, 8 weeks of each treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil Once a Day [T(OaD)] | Sildenafil as Needed [S(PRN)] | Tadalafil as Needed [T(PRN)]
Number analyzed (Participants) | 350 | 348 | 355
units on a scale
  Baseline | 15.60 (6.26) | 15.40 (6.27) | 15.55 (6.23)
  Change from Baseline | 8.68 (6.94) | 9.70 (7.01) | 9.54 (7.00)
Statistical Analysis 1: Comparison: Tadalafil Once a Day [T(OaD)] vs Sildenafil as Needed [S(PRN)]; Test type: Superiority or Other; p = 0.004, t-test — p-value is for the difference between Tadalafil OaD and Sildenafil PRN Change from Baseline in LS Means; Kenward-Roger approximation was used for denominator degrees of freedom in the mixed model; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-1.43 to -0.27], Standard Error of Mean 0.30
Statistical Analysis 2: Comparison: Tadalafil Once a Day [T(OaD)] vs Tadalafil as Needed [T(PRN)]; Test type: Superiority or Other; p = 0.007, t-test — p-value is for the difference between Tadalafil OaD and Tadalafil PRN Change from Baseline in LS Means; Kenward-Roger approximation was used for denominator degrees of freedom in the mixed model; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-1.37 to -0.22], Standard Error of Mean 0.29

6. Secondary Outcome: Change From Baseline to Endpoint in the Proportion of Days With at Least One Morning Erection
Time Frame: baseline, 8 weeks of each treatment
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Tadalafil Once a Day [T(OaD)] | Tadalafil as Needed [T(PRN)] | Sildenafil as Needed [S(PRN)]
Number analyzed (Participants) | 352 | 355 | 347
proportion of days
  Baseline | 0.28 (0.26) | 0.28 (0.26) | 0.27 (0.26)
  Change from Baseline | 0.26 (0.29) | 0.20 (0.25) | 0.11 (0.24)
Statistical Analysis 1: Comparison: Tadalafil Once a Day [T(OaD)] vs Tadalafil as Needed [T(PRN)]; Test type: Superiority or Other; p < 0.001, t-test — p-value is for difference between Tadalafil OaD and Tadalafil PRN Change from Baseline in LS Means; Kenward-Roger approximation was used for denominator degrees of freedom in the mixed model; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [0.03 to 0.09], Standard Error of Mean 0.01
Statistical Analysis 2: Comparison: Tadalafil Once a Day [T(OaD)] vs Sildenafil as Needed [S(PRN)]; Test type: Superiority or Other; p < 0.001, t-test — p-value is for difference between Tadalafil OaD and Sildenafil PRN Change from Baseline in LS Means; Kenward-Roger approximation was used for denominator degrees of freedom in the mixed model; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [0.06 to 0.12], Standard Error of Mean 0.01

7. Secondary Outcome: Change From Baseline to Endpoint in the Intercourse Satisfaction (IS) Domain of the IIEF
Description: Self-reported intercourse satisfaction over the past 4 weeks. Scores range from 0 (low/no satisfaction to 5 (high satisfaction), thus the 3 questions of the IIEF-IS domain range from 0 to 15.
Time Frame: baseline, 8 weeks of each treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil Once a Day [T(OaD)] | Sildenafil as Needed [S(PRN)] | Tadalafil as Needed [T(PRN)]
Number analyzed (Participants) | 350 | 348 | 355
units on a scale
  Baseline | 8.35 (2.76) | 8.34 (2.77) | 8.37 (2.73)
  Change from Baseline | 3.33 (3.16) | 3.99 (3.17) | 3.83 (3.13)
Statistical Analysis 1: Comparison: Tadalafil Once a Day [T(OaD)] vs Sildenafil as Needed [S(PRN)]; Test type: Superiority or Other; p < 0.001, t-test — p-value is for difference between Tadalafil OaD and Sildenafil PRN Change from Baseline in LS Means; Kenward-Roger approximation was used for denominator degrees of freedom in the mixed model; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-0.91 to -0.36], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Tadalafil Once a Day [T(OaD)] vs Tadalafil as Needed [T(PRN)]; Test type: Superiority or Other; p < 0.001, t-test — p-value is for difference between Tadalafil OaD and Tadalafil PRN Change from Baseline in LS Means; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-0.78 to -0.23], Standard Error of Mean 0.14

8. Secondary Outcome: Change From Baseline to Endpoint in the Overall Satisfaction (OS) Domain of the IIEF
Description: Self-reported overall satisfaction over the past 4 weeks. Scores range from 0 (low/no satisfaction to 5 (high satisfaction), thus the 2 questions of the IIEF-OS domain range from 0 to 10.
Time Frame: baseline, 8 weeks of each treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil Once a Day [T(OaD)] | Sildenafil as Needed [S(PRN)] | Tadalafil as Needed [T(PRN)]
Number analyzed (Participants) | 350 | 348 | 355
units on a scale
  Baseline | 5.26 (2.34) | 5.22 (2.36) | 5.27 (2.34)
  Change from Baseline | 2.60 (2.61) | 2.87 (2.55) | 2.84 (2.58)
Statistical Analysis 1: Comparison: Tadalafil Once a Day [T(OaD)] vs Sildenafil as Needed [S(PRN)]; Test type: Superiority or Other; p = 0.055, t-test — p-value is for the difference between Tadalafil OaD and Sildenafil PRN Change from Baseline in LS Means; Kenward-Roger approximation was used for denominator degrees of freedom in the mixed model; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.44 to 0.00], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Tadalafil Once a Day [T(OaD)] vs Tadalafil as Needed [T(PRN)]; Test type: Superiority or Other; p = 0.046, t-test — p-value is for the difference between Tadalafil OaD and Tadalafil PRN Change from Baseline in LS Means; Kenward-Roger approximation was used for denominator degrees of freedom in the mixed model; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.44 to 0.00], Standard Error of Mean 0.11

9. Secondary Outcome: Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) Score at Endpoint
Description: EDITS is a questionnaire-based inventory capturing a participant's subjective evaluation of treatment for the participant's erection problems. All items on the 11-item Patient EDITS were scored from zero (no satisfaction or dissatisfaction) to four (high satisfaction). The EDITS Summary Score (transformed) is obtained by adding each individual score for all questions, dividing by the number of questions, and multiplying by 25, so that EDITS scores could range from a low of 0 (extremely low treatment satisfaction) to a high of 100 (extremely high treatment satisfaction).
Time Frame: 8 weeks of each treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil Once a Day [T(OaD)] | Sildenafil as Needed [S(PRN)] | Tadalafil as Needed [T(PRN)]
Number analyzed (Participants) | 351 | 348 | 355
units on a scale | 75.81 (22.36) | 75.68 (19.58) | 79.50 (19.56)
Statistical Analysis 1: Comparison: Tadalafil Once a Day [T(OaD)] vs Sildenafil as Needed [S(PRN)]; Test type: Superiority or Other; p = 0.004, t-test — p-value is for the difference between Tadalafil PRN and Sildenafil PRN change in LS Means; Kenward-Roger approximation was used for denominator degrees of freedom in the mixed model; Mean Difference (Final Values) = 3.66, 95% CI 2-sided [1.16 to 6.17], Standard Error of Mean 1.27
Statistical Analysis 2: Comparison: Tadalafil Once a Day [T(OaD)] vs Tadalafil as Needed [T(PRN)]; Test type: Superiority or Other; p = 0.006, t-test — p-value is for the difference between Tadalafil OaD and Tadalafil PRN change in LS Means; Kenward-Roger approximation was used for denominator degrees of freedom in the mixed model; Mean Difference (Final Values) = -3.55, 95% CI 2-sided [-6.05 to -1.04], Standard Error of Mean 1.27

10. Secondary Outcome: Number of Participants With at Least One Serious Adverse Event
Description: Serious adverse events are listed in the Reported Adverse Event module.
Time Frame: baseline through 26 weeks (including two washout periods of 1 week each)
Measure: Number; unit: participants
Arm/Group | Tadalafil Once a Day [T(OaD)] | Sildenafil as Needed [S(PRN)] | Tadalafil as Needed [T(PRN)]
Number analyzed (Participants) | 378 | 378 | 378
participants | 4 | 5 | 2

11. Secondary Outcome: Change From Baseline to Endpoint in the Self-Esteem And Relationship (SEAR) Questionnaire Transformed Total Score
Description: Measures improvement in self-esteem and relationship satisfaction. Questionnaire consists of two domains, Sexual Relationship (items 1-8) and Confidence (items 9-14). Overall score is transformed onto a 0 (least favorable) to 100 (most favorable) scale. Overall score was calculated from two domains and subscales scores.
Time Frame: baseline, 8 weeks of each treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil Once a Day [T(OaD)] | Sildenafil as Needed [S(PRN)] | Tadalafil as Needed [T(PRN)]
Number analyzed (Participants) | 348 | 347 | 355
units on a scale
  Baseline | 50.28 (21.36) | 50.50 (21.58) | 50.69 (21.32)
  Change from Baseline | 22.94 (24.86) | 22.87 (24.43) | 24.13 (24.53)
Statistical Analysis 1: Comparison: Tadalafil Once a Day [T(OaD)] vs Sildenafil as Needed [S(PRN)]; Test type: Superiority or Other; p = 0.915, t-test — p-value is for the difference between Tadalafil OaD and Sildenafil PRN Change from Baseline in LS Means; Kenward-Roger approximation was used for denominator degrees of freedom in the mixed model; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-1.95 to 2.17], Standard Error of Mean 1.05
Statistical Analysis 2: Comparison: Tadalafil Once a Day [T(OaD)] vs Tadalafil as Needed [T(PRN)]; Test type: Superiority or Other; p = 0.212, t-test — p-value is for the difference between Tadalafil OaD and Tadalafil PRN Change from Baseline in LS Means; Kenward-Roger approximation was used for denominator degrees of freedom in the mixed model; Mean Difference (Final Values) = -1.30, 95% CI 2-sided [-3.35 to 0.74], Standard Error of Mean 1.04

12. Secondary Outcome: Question 1 "I Felt as if I Did Not Have ED" Score of the Patient Perception and Feelings Questions (PPF-Q) at Endpoint
Description: Scores for Question 1 range from 0 (not at all) to 4 (extremely).
Time Frame: 8 weeks of each treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil Once a Day [T(OaD)] | Sildenafil as Needed [S(PRN)] | Tadalafil as Needed [T(PRN)]
Number analyzed (Participants) | 349 | 348 | 355
units on a scale | 1.83 (1.25) | 1.78 (1.13) | 1.77 (1.22)
Statistical Analysis 1: Comparison: Tadalafil Once a Day [T(OaD)] vs Sildenafil as Needed [S(PRN)]; Test type: Superiority or Other; p = 0.403, Generalized Linear Mixed Model — p-value is for the difference between Tadalafil OaD and Sildenafil PRN in LS Means; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.09 to 0.22], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Tadalafil Once a Day [T(OaD)] vs Tadalafil as Needed [T(PRN)]; Test type: Superiority or Other; p = 0.367, Generalized Linear Mixed Model — p-value is for the difference between Tadalafil OaD and Tadalafil PRN in LS Means; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.08 to 0.23], Standard Error of Mean 0.08

13. Secondary Outcome: Question 2 "I Felt in Control of my Sex Life" Score of the Patient Perception and Feelings Questions (PPF-Q) at Endpoint
Description: Scores for Question 2 range from 0 (not at all) to 4 (extremely).
Time Frame: 8 weeks of each treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil Once a Day [T(OaD)] | Sildenafil as Needed [S(PRN)] | Tadalafil as Needed [T(PRN)]
Number analyzed (Participants) | 349 | 348 | 355
units on a scale | 2.33 (1.09) | 2.14 (1.01) | 2.36 (1.10)
Statistical Analysis 1: Comparison: Tadalafil Once a Day [T(OaD)] vs Sildenafil as Needed [S(PRN)]; Test type: Superiority or Other; p = 0.002, Generalized Linear Mixed Model — p-value is for the difference between Tadalafil OaD and Sildenafil PRN in LS Means; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [0.07 to 0.32], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Tadalafil Once a Day [T(OaD)] vs Tadalafil as Needed [T(PRN)]; Test type: Superiority or Other; p = 0.722, Generalized Linear Mixed Model — p-value is for the difference between Tadalafil OaD and Tadalafil PRN in LS Means; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.15 to 0.10], Standard Error of Mean 0.06

14. Secondary Outcome: Question 3 "I Felt the Drug Was in Control of my Erections" Score of the Patient Perception and Feelings Questions (PPF-Q) at Endpoint
Description: Scores for Question 3 range from 0 (not at all) to 4 (extremely).
Time Frame: 8 weeks of each treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil Once a Day [T(OaD)] | Sildenafil as Needed [S(PRN)] | Tadalafil as Needed [T(PRN)]
Number analyzed (Participants) | 349 | 348 | 355
units on a scale | 1.99 (1.19) | 2.28 (1.12) | 2.50 (1.14)
Statistical Analysis 1: Comparison: Tadalafil Once a Day [T(OaD)] vs Sildenafil as Needed [S(PRN)]; Test type: Superiority or Other; p < 0.001, Generalized Linear Mixed Model — p-value is for the difference between Tadalafil OaD and Sildenafil PRN in LS Means; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-0.65 to -0.37], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Tadalafil Once a Day [T(OaD)] vs Tadalafil as Needed [T(PRN)]; Test type: Superiority or Other; p < 0.001, Generalized Linear Mixed Model — p-value is for the difference between Tadalafil OaD and Tadalafil PRN in LS Means; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.43 to -0.16], Standard Error of Mean 0.07

15. Secondary Outcome: Question 4 "I Felt Like a Whole Man" Score of the Patient Perception and Feelings Questions (PPF-Q) at Endpoint
Description: Scores for Question 4 range from 0 (not at all) to 4 (extremely).
Time Frame: 8 weeks of each treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil Once a Day [T(OaD)] | Sildenafil as Needed [S(PRN)] | Tadalafil as Needed [T(PRN)]
Number analyzed (Participants) | 349 | 348 | 355
units on a scale | 2.53 (1.10) | 2.57 (1.06) | 2.44 (0.99)
Statistical Analysis 1: Comparison: Tadalafil Once a Day [T(OaD)] vs Sildenafil as Needed [S(PRN)]; Test type: Superiority or Other; p = 0.070, Generalized Linear Mixed Model — p-value is for the difference between Tadalafil OaD and Sildenafil PRN in LS Means; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.01 to 0.22], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Tadalafil Once a Day [T(OaD)] vs Tadalafil as Needed [T(PRN)]; Test type: Superiority or Other; p = 0.637, Generalized Linear Mixed Model — p-value is for the difference between Tadalafil OaD and Tadalafil PRN in LS Means; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.14 to 0.09], Standard Error of Mean 0.06

ADVERSE EVENTS:
Groups:
- Sildenafil Citrate as Needed [S(PRN)]: Sildenafil citrate 100 mg as needed [S(PRN)]
Arm/Group | Tadalafil Once a Day [T(OaD)] | Sildenafil Citrate as Needed [S(PRN)] | Tadalafil as Needed [T(PRN)]
Serious Adverse Events (participants affected / at risk) | 4/378 | 5/378 | 2/378
Other Adverse Events (participants affected / at risk) | 66/378 | 73/378 | 70/378
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil Once a Day [T(OaD)] (N=378) | Sildenafil Citrate as Needed [S(PRN)] (N=378) | Tadalafil as Needed [T(PRN)] (N=378)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Elbow operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil Once a Day [T(OaD)] (N=378) | Sildenafil Citrate as Needed [S(PRN)] (N=378) | Tadalafil as Needed [T(PRN)] (N=378)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypogonadism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 2 (2) | 2 (2)
Abnormal sensation in eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Cyanopsia (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Metamorphopsia (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Visual brightness (Eye disorders) | 0 (0) | 1 (10) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (6) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 5 (15) | 4 (7)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 3 (9) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (10) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Ear infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3) | 5 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (19) | 0 (0)
Headache (Nervous system disorders) | 10 (10) | 13 (20) | 8 (18)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Balanitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Ejaculation failure (Reproductive system and breast disorders) | 0 (0) | 1 (4) | 2 (2)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Priapism (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (15) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (2) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 6 (6) | 8 (26) | 3 (3)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days